CLINICAL TRIAL: NCT00307671
Title: Treatment of Necrotizing Vasculitides for Patients Older Than 65 Years Comparison of Two Strategies Combining Steroids With or Without Immunosuppressants
Brief Title: Treatment of Necrotizing Vasculitides for Patients Older Than 65 Years
Acronym: CORTAGE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P040425
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2007-03

CONDITIONS: Vasculitis; Wegener's Granulomatosis; Microscopic Polyangiitis; Churg-Strauss Syndrome; Polyarteritis Nodosa
Keywords: Systemic necrotizing vasculitides; corticosteroids; azathioprine; mycophenolate mofetil;; cyclophosphamide; Elderly patients; Randomized controlled trial
MeSH Terms: conditions — Vasculitis; Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Churg-Strauss Syndrome; Polyarteritis Nodosa | interventions — Prednisone; Methylprednisolone; Cyclophosphamide; Azathioprine; Mycophenolic Acid; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Other): conventional treatment
  Interventions: Drug: prednisone, methylprednisolone,cyclophosphamides; Drug: Mycophenolate mofetil,methotrexate
- B (Experimental): reduction dose
  Interventions: Drug: Cyclophosphamide, Azathioprine,prednisone,methylprednisolone; Drug: Mycophenolate mofetil,methotrexate

INTERVENTIONS:
Drug: prednisone, methylprednisolone,cyclophosphamides — treatment conventional
  Arms: A
Drug: Cyclophosphamide, Azathioprine,prednisone,methylprednisolone — reduction dose
  Arms: B
Drug: Mycophenolate mofetil,methotrexate — in the treatment conventional and in the reduction dose

SUMMARY:
The aim of this trial is to lower the morbidity rate in elderly patients affected with systemic necrotizing vasculitides, by reducing mortality and improving global outcome.

DETAILED DESCRIPTION:
Systemic necrotizing vasculitides are severe diseases associated with a high mortality rate in elderly.

Although corticosteroids and immunosuppressants are effective, they can induce some side-effects, especially in this latter patients.

Preliminary data indicate that systemic necrotizing vasculitides (SNV) occurring in patients over 65 years have a poorer outcome than in younger patients (mortality rate of 76 % vs. 69 % at 5 years, respectively) and that 68,4 % of the elderly experience treatment side-effects.

In this trial, patients will be randomly assigned to receive either low doses of corticosteroids systematically in combination with immunosuppressants (CYC then azathioprine) or usual regimen with corticosteroids combined with immunosuppressants only if factor(s) of poor prognosis is present (this latter regimen relying on previously published therapeutic guidelines).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed WG, MPA, PAN without HBV infection, or CSS
* Patients can be still be enrolled within 1 month after starting corticosteroids if prescribed according to protocol.
* within or after the 65th of anniversary
* Age ≥ 65 years

Exclusion Criteria:

* Any cytotoxic drug within previous year
* Co-existence of another systemic autoimmune disease, e.g., SLE, RA
* Virus-associated vasculitides
* HIV positivity
* Malignancy (usually excluded unless approved by the trial coordinator)
* Age < 65 years
* Inability to give informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 108 (Actual)
Dates: Start 2005-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Number of side effects (morbidity) | at 3 years

SECONDARY OUTCOMES:
Survival | at 3 years
Efficacy of treatment (remission rate) | during the 3 years
Relapse rate | at 3 years
Cumulative dose exposure to OCS and AZA | at 3 years
Cumulative BVAS (AUC), VDI, HAQ-DI, SF-36 values | at 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Loïc Guillevin, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, Paris, France

REFERENCES:
- [Derived] Pagnoux C, Quemeneur T, Ninet J, Diot E, Kyndt X, de Wazieres B, Reny JL, Puechal X, le Berruyer PY, Lidove O, Vanhille P, Godmer P, Fain O, Blockmans D, Bienvenu B, Rollot F, Ait el Ghaz-Poignant S, Mahr A, Cohen P, Mouthon L, Perrodeau E, Ravaud P, Guillevin L; French Vasculitis Study Group. Treatment of systemic necrotizing vasculitides in patients aged sixty-five years or older: results of a multicenter, open-label, randomized controlled trial of corticosteroid and cyclophosphamide-based induction therapy. Arthritis Rheumatol. 2015 Apr;67(4):1117-27. doi: 10.1002/art.39011. PMID 25693055